CLINICAL TRIAL: NCT00438399
Title: Subject Preference Comparison Between Clobetasol Propionate Shampoo, 0.05% and Three Other Topical Corticosteroids in the Treatment of Moderate to Severe Scalp Psoriasis
Brief Title: Subject Preference for Scalp Psoriasis Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29064; 2006-003073-27 (EudraCT Number)
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-11

CONDITIONS: Scalp Psoriasis
Keywords: 1 Galderma,; 2 Scalp Psoriasis; 3 Subject preference; 4 Clobetasol propionate; 5 Shampoo

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- C. propionate-Wash out-Corticosteroid 1 (Active Comparator): Clobetasol propionate Shampoo:
  * Dose or Concentration: Clobetasol propionate 0.05% shampoo
  * Mode and Frequency of Administration: Topical Once daily to the dry scalp, to be lathered and rinsed after 15 minutes
  * Duration of Treatment: 4 weeks as a maximum
  Wash-out up to 8 weeks
  Corticosteroid 1:
  * Dose or Concentration: Corticosteroid 1 Foam
  * Mode and Frequency of Administration:Twice daily, a "golf-ball" sized amount to be massaged into the affected area of the scalp
  * Duration of Treatment: 4 weeks as a maximum
  Interventions: Drug: C. propionate - Corticosteroid 1
- C. propionate-Wash out-Corticosteroid 2 (Active Comparator): Clobetasol propionate Shampoo:
  * Dose or Concentration: Clobetasol propionate 0.05% shampoo
  * Mode and Frequency of Administration: Topical Once daily to the dry scalp, to be lathered and rinsed after 15 minutes
  * Duration of Treatment: 4 weeks as a maximum
  Corticosteroid 2:
  * Dose or Concentration: Corticosteroid 2 Lotion
  * Mode and Frequency of Administration: Twice daily, a thin film to be applied to the affected area of the scalp and massaged gently and thoroughly into the skin
  * Duration of Treatment: 4 weeks as a maximum
  Interventions: Drug: C. propionate- Corticosteroid 2
- C. propionate-Wash out-Corticosteroid 3 (Active Comparator): Clobetasol propionate Shampoo:
  * Dose or Concentration: Clobetasol propionate 0.05% shampoo
  * Mode and Frequency of Administration: Topical Once daily to the dry scalp, to be lathered and rinsed after 15 minutes
  * Duration of Treatment: 4 weeks as a maximum
  Corticosteroid 3:
  * Dose or Concentration: Corticosteroid 3 Scalp application
  * Mode and Frequency of Administration: Twice daily, a thin film to be applied into the affected area of the dry scalp and rubbed gently into the scalp
  * Duration of Treatment: 4 weeks as a maximum
  Interventions: Drug: C. propionate -Corticosteroid 3
- Corticosteroid 1-Wash out-C. propionate (Active Comparator): Clobetasol propionate Shampoo:
  * Dose or Concentration: Clobetasol propionate 0.05% shampoo
  * Mode and Frequency of Administration: Topical Once daily to the dry scalp, to be lathered and rinsed after 15 minutes
  * Duration of Treatment: 4 weeks as a maximum
  Corticosteroid 1:
  * Dose or Concentration: Corticosteroid 1 Foam
  * Mode and Frequency of Administration:Twice daily, a "golf-ball" sized amount to be massaged into the affected area of the scalp
  * Duration of Treatment: 4 weeks as a maximum
  Interventions: Drug: Corticosteroid 1- C. propionate
- Corticosteroid 2-Wash out-C. propionate (Active Comparator): Clobetasol propionate Shampoo:
  * Dose or Concentration: Clobetasol propionate 0.05% shampoo
  * Mode and Frequency of Administration: Topical Once daily to the dry scalp, to be lathered and rinsed after 15 minutes
  * Duration of Treatment: 4 weeks as a maximum
  Corticosteroid 2:
  * Dose or Concentration: Corticosteroid 2 Lotion
  * Mode and Frequency of Administration: Twice daily, a thin film to be applied to the affected area of the scalp and massaged gently and thoroughly into the skin
  * Duration of Treatment: 4 weeks as a maximum
  Interventions: Drug: Corticosteroid 2 - C. propionate
- Corticosteroid 3-Wash out-C. propionate (Active Comparator): Clobetasol propionate Shampoo:
  * Dose or Concentration: Clobetasol propionate 0.05% shampoo
  * Mode and Frequency of Administration: Topical Once daily to the dry scalp, to be lathered and rinsed after 15 minutes
  * Duration of Treatment: 4 weeks as a maximum
  Corticosteroid 3:
  * Dose or Concentration: Corticosteroid 3 Scalp application
  * Mode and Frequency of Administration: Twice daily, a thin film to be applied into the affected area of the dry scalp and rubbed gently into the scalp
  * Duration of Treatment: 4 weeks as a maximum
  Interventions: Drug: Corticosteroid 3 - C. propionate

INTERVENTIONS:
Drug: C. propionate - Corticosteroid 1 — Twice daily application
  Other Names: CP shampoo compared to Corticosteroid 1
  Arms: C. propionate-Wash out-Corticosteroid 1
Drug: C. propionate- Corticosteroid 2 — Twice daily application
  Other Names: CP Shampoo compared to Corticosteroid 2
  Arms: C. propionate-Wash out-Corticosteroid 2
Drug: C. propionate -Corticosteroid 3 — Twice daily application
  Other Names: CP Shampoo compared to Corticosteroid 3
  Arms: C. propionate-Wash out-Corticosteroid 3
Drug: Corticosteroid 1- C. propionate — Twice daily application
  Other Names: Corticosteroid 1 compared to CP Shampoo
  Arms: Corticosteroid 1-Wash out-C. propionate
Drug: Corticosteroid 2 - C. propionate — Twice daily application
  Other Names: Corticosteroid 2 compared to CP Shampoo
  Arms: Corticosteroid 2-Wash out-C. propionate
Drug: Corticosteroid 3 - C. propionate — Twice daily application
  Other Names: Corticosteroid 3 compared to CP Shampoo
  Arms: Corticosteroid 3-Wash out-C. propionate

SUMMARY:
The scalp is one of the most common affected sites in psoriatic patients as 79% of them have scalp involvement.It has also a psychological aspect with 31% of patients with scalp psoriasis indicating distress.

Topical agents remain the mainstay of treatment for scalp psoriasis. However, they are not always ideal because they might be inconvenient and messy to use, stain or damage hair.

The test shampoo, Clobetasol propionate Shampoo 0.05% (marketed in the USA under the tradename of Clobex®) was developed to provide the strongest available corticosteroid as a short-contact therapy in order to improve the chances of it being effective and reduce the potential for traditional side-effects.

The objective of this study is to compare subject's overall preference between Clobetasol propionate shampoo 0.05% and three other topical corticosteroids in the treatment of moderate to severe scalp psoriasis.

DETAILED DESCRIPTION:
This study will be a multi-centre, investigator blinded, randomized, cross-over, intra-individual comparison in three parallel groups.

In each parallel group, Clobetasol propionate shampoo, 0.05% will be compared to one of the three chosen competitors, following a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older,
* Subjects with moderate to severe scalp psoriasis,
* Subjects who signed written informed consent prior to any study procedures.

Exclusion Criteria:

* Subjects who need systemic treatment for their body psoriasis,
* Subjects who are at risk in terms of precautions, warnings and contra-indication,
* Female subjects who are pregnant, nursing or planning a pregnancy during the study,
* Subjects with a specific washout period for topical treatment(s) on the scalp,
* Subjects with a specific washout period for systemic treatment(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Giannetti, Professor, Principal Investigator — Clinica Dermatologica Azienda Ospedaliera Policinico di Modena - Italy
Locations (1):
- Clinica Dermatologica Azienda Ospedaliera Policlinico di Modena, Modena, Italy

REFERENCES:
- See also: Study product information — http://www.clobex.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in 18 centres in Italy, Spain, United Kingdom and Germany between 19 February 2007 until 22 January 2008
Pre-assignment Details: 219 participants recruited.
Groups:
- C. Propionate-Wash Out-Corticosteroid 1: Clobetasol propionate Shampoo first, then Corticosteroid 1
- Corticosteroid 1-Wash Out-C. Propionate: Corticosteroid 1 first then Clobetasol propionate Shampoo
- C. Propionate-Wash Out-Corticosteroid 2: Clobetasol propionate Shampoo first, then Corticosteroid 2
- Corticosteroid 2-Wash Out-C. Propionate: Corticosteroid 2 first, then Clobetasol propionate shampoo
- C. Propionate -Wash Out-Corticosteroid 3: Clobetasol propionate shampoo first then Corticosteroid 3
- Corticosteroid 3-Wash Out-C. Propionate: Corticosteroid 3 first, then Clobetasol propionate
Period: Overall Study
Arm/Group | C. Propionate-Wash Out-Corticosteroid 1 | Corticosteroid 1-Wash Out-C. Propionate | C. Propionate-Wash Out-Corticosteroid 2 | Corticosteroid 2-Wash Out-C. Propionate | C. Propionate -Wash Out-Corticosteroid 3 | Corticosteroid 3-Wash Out-C. Propionate
Started | 38 | 40 | 35 | 36 | 33 | 37
TREATED & ANALYZED | 30 | 32 | 28 | 32 | 30 | 31
Completed | 30 | 32 | 28 | 32 | 30 | 31
Not Completed | 8 | 8 | 7 | 4 | 3 | 6
Not completed — Lost to Follow-up | 2 | 2 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 6 | 3 | 2 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Subje stopped study | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Patien stopped study at visit 4 by error | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- C. Propionate Compared to Corticosteroid 1: C. propionate shampoo: once daily Corticosteroid 1 foam:twice daily
- C. Propionate Compared to Corticosteroid 2: C. propionate shampoo: once daily Corticosteroid 2 lotion: twice daily
- C. Propionate Compared to Corticosteroid 3: C. propionate shampoo: once daily Corticosteroid 3 scalp application: twice daily
- Total: Total of all reporting groups
Arm/Group | C. Propionate Compared to Corticosteroid 1 | C. Propionate Compared to Corticosteroid 2 | C. Propionate Compared to Corticosteroid 3 | Total
Number analyzed (Participants) | 78 | 71 | 70 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 58 | 55 | 57 | 170
  >=65 years | 20 | 15 | 13 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (15.9) | 49.2 (14.9) | 47.8 (16.2) | 49.3 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 32 | 36 | 113
  Male | 33 | 39 | 34 | 106
Region of Enrollment [Number; unit: participants]
  Italy | 16 | 16 | 16 | 48
  United Kingdom | 17 | 15 | 11 | 43
  Spain | 9 | 5 | 9 | 23
  Germany | 36 | 35 | 34 | 105

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Preffering Clobetasol Propionate Shampoo Better Than Comparator
Description: Subjects' Overall preference at the end of Period II. The purpose was to demonstrate a superiority of Clobetasol propionate shampoo 0.05% therapy compared to any of three other topical comparators, in terms of subject's overall preference: "C. propionate shampoo a lot better than the comparator",C. propionate shampoo a lillte bit better than the comparator", "Comparator a lot better than C. propionate shampoo", Comparator a lillte bit better than C. propionate shampoo". This was to be shown using a non parametric two-sided Wilcoxon rank Signed test, on Intention to Treat (ITT) population.
Time Frame: End of period II (up to 16 weeks)
Population: Intent to Treat population (ITT).
Measure: Number; unit: Percentage of participants
Arm/Group | C. Propionate Compared to Corticosteroid 1 | C. Propionate Compared to Corticosteroid 2 | C. Propionate Compared to Corticosteroid 3
Number analyzed (Participants) | 63 | 60 | 55
Percentage of participants | 28.5 | 31.6 | 21.8
Statistical Analysis 1: Comparison: C. Propionate Compared to Corticosteroid 1; The purpose of the study was to demonstrate the superiority of Clobetasol propionate shampoo over one of three other comparators, in terms of Subject's overall preference. It was to be analyzed using a non parametric two-sided Wilcoxon rank Signed test on ITT population; Test type: Superiority or Other; p = 0.0003, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: C. Propionate Compared to Corticosteroid 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: C. Propionate Compared to Corticosteroid 3; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the study period (maximum of 16 weeks)
Groups:
- Corticosteroid 1: All subjects having used Corticosteroid 1
- Corticosteroid 2: All subjects having used Corticosteroid 2
- Corticosteroid 3: All subjects having used Corticosteroid 3
- Clobetasol Propionate Shampoo: All subjects having used Clobetasol propionate shampoo
Arm/Group | Corticosteroid 1 | Corticosteroid 2 | Corticosteroid 3 | Clobetasol Propionate Shampoo
Serious Adverse Events (participants affected / at risk) | 0/72 | 2/67 | 1/65 | 3/199
Other Adverse Events (participants affected / at risk) | 5/72 | 11/67 | 20/65 | 5/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroid 1 (N=72) | Corticosteroid 2 (N=67) | Corticosteroid 3 (N=65) | Clobetasol Propionate Shampoo (N=199)
UNCLEAR ABDOMINAL PAIN - MECHANICAL SUBILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HOSPITALISATION DUE TO NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HOSPITALIZATION DUE TO MALAISE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTOLITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroid 1 (N=72) | Corticosteroid 2 (N=67) | Corticosteroid 3 (N=65) | Clobetasol Propionate Shampoo (N=199)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
HORDEOLUM (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 3 (4) | 3 (3) | 0 (0)
FOLLICULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
SKIN BURNING SENSATION (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IMPETIGO (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EXPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor to review and approval at least 2 months prior to the date of intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.